CLINICAL TRIAL: NCT03959189
Title: Double-Blind, Placebo-Controlled, Dose-Range-Finding, Crossover Trial of Single Day Administration of ERX-963 in Adults With Myotonic Dystrophy Type 1
Brief Title: Safety, Tolerability and Pharmacokinetics of ERX-963 in Adults With Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Expansion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ERX-963-001
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-05

CONDITIONS: Myotonic Dystrophy, Type 1 (DM1); Myotonic Dystrophy
Keywords: Excessive Daytime Sleepiness; hypersomnia
MeSH Terms: conditions — Myotonic Dystrophy; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ERX-963 then placebo (Experimental): Participants in this arm will receive ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
  Interventions: Drug: ERX-963
- Placebo then ERX-963 (Experimental): Participants in this arm will receive placebo followed by a washout period. After the washout period, participants will receive ERX-963.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ERX-963 — Active medicine
  Arms: ERX-963 then placebo
Drug: Placebo — Comparator
  Arms: Placebo then ERX-963

SUMMARY:
Participants in this study will receive two treatments, placebo and ERX-963, on different days in a randomized fashion.

The primary purpose of this study is to investigate the safety and tolerability of ERX-963 in participants diagnosed with Myotonic Dystrophy, Type 1 (DM1).

The secondary purpose is to evaluate the potential of ERX-963 treatment to reduce excessive daytime sleepiness / hypersomnia and improve cognitive function in DM1 participants compared to placebo treatment.

DETAILED DESCRIPTION:
This study is evaluating single administration of two dose levels of ERX-963 to explore the relationship between dose, safety, tolerability, exposure and clinical benefit. This is a multi-center, randomized, double-blind, placebo-controlled, two-treatment period crossover study in two cohorts of participants with DM1.

Participants who have consented and meet eligibility criteria will receive two treatments, placebo and ERX-963, in a randomized crossover fashion with a washout period between the treatments. On treatment days, participants will receive treatment followed by repeated blood collection for pharmacokinetic analysis and administration of a battery of outcome measures relevant to sleep and cognition.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 65 years of age
* DM1 defined by genetic testing or clinical-confirmation
* Epworth Sleepiness Scale (ESS) of > 11 or participants who have long sleep periods of an average of > 10 hours a day
* Age of onset of DM1 greater than 16 years

Key Exclusion Criteria:

* Significant respiratory compromise
* Significant cardiac disease
* Diagnosis of symptomatic Restless Leg Syndrome or significant untreated nocturnal hypoxias
* Significant moderate to severe hepatic insufficiency
* Clinically active depression, anxiety, or other medical condition that, in the investigator's opinion, would interfere with the safety and efficacy assessments
* History of seizures
* History of panic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Ehrich, MD, Study Director — Chief Medical Officer
Locations (4):
- United States (4):
  - Stanford Neurosciences Health Center, Palo Alto, California
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Expansion Therapeutics Corporate Website — https://www.expansionrx.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2019 and March 2020, 12 patients were enrolled and treated with ERX-963 at three sites in the United States (Stanford University Neurosciences Health Center, University of Iowa Hospitals and Clinics, and Sleep Specialists of South Florida).
Groups:
- Cohort 1: 1 mg ERX-963: Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 1 mg of ERX-963.
  Sequence 2: Participants will receive 1 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
- Cohort 2: 2 mg ERX-963: Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 2 mg of ERX-963.
  Sequence 2: Participants will receive 2 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
Period: Overall Study
Arm/Group | Cohort 1: 1 mg ERX-963 | Cohort 2: 2 mg ERX-963
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 1 mg ERX-963 | Cohort 2: 2 mg ERX-963 | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Median (Full Range); unit: years] | 54.0 [47 to 59] | 44.0 [29 to 56] | 51.5 [29 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events, Serious Adverse Events, and Drug-related Adverse Events [Safety and Tolerability] After a Single Dose of ERX-963 vs. Placebo
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. Treatment-emergent AEs were AEs which started between the date and time of study drug dosing and through Study Day 2, within each period. Drug-related AEs were assessed by the investigator to determine the relationship (related or unrelated) between the study intervention and each AE occurrence.
Time Frame: Adverse Events were collected from screening to the End of Study Visit, up to 57 days
Population: The safety population is defined as all participants who sign the study-specific informed consent documents and received at least 1 dose of ERX-963 or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 1 mg ERX-963: The crossover design tests each subject under different treatment conditions allowing for each subject to serve as their own control.
  Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 1 mg of ERX-963.
  Sequence 2: Participants will receive 1 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
- Cohort 2: 2 mg ERX-963: The crossover design tests each subject under different treatment conditions allowing for each subject to serve as their own control.
  Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 2 mg of ERX-963.
  Sequence 2: Participants will receive 2 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
Arm/Group | Cohort 1: 1 mg ERX-963 | Cohort 2: 2 mg ERX-963
Number analyzed (Participants) | 7 | 5
Participants
  Serious Adverse Events | 0 | 0
  Drug-related AEs in Placebo period | 1 | 1
  Drug-related AEs in ERX-963 period | 0 | 0
  TEAEs in Placebo period | 0 | 2
  TEAEs in ERX-963 period | 1 | 1

2. Secondary Outcome: Assess the Effect of ERX-963 on the Stanford Sleepiness Scale Score Compared to the Effect of Placebo
Description: Participants will self-report their level of sleepiness by self-rated questionnaire "Stanford Sleepiness Scale" (SSS). This is a single item questionnaire on a 7-point scale (1-7). Higher values indicate worse outcome.
Time Frame: From dosing to approximately 2 hours
Population: All treated participants who completed all the protocol specified assessments in both treatment periods were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort 1: Placebo Period; Cohort 2: Placebo Period; Cohort 2: 2 mg ERX-963 Period: The crossover design tests each subject under different treatment conditions allowing for each subject to serve as their own control.
  Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 2 mg of ERX-963.
  Sequence 2: Participants will receive 2 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
- Cohort 1: 1 mg ERX-963 Period: The crossover design tests each subject under different treatment conditions allowing for each subject to serve as their own control.
  Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 1 mg of ERX-963.
  Sequence 2: Participants will receive 1 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
Arm/Group | Cohort 1: Placebo Period | Cohort 1: 1 mg ERX-963 Period | Cohort 2: Placebo Period | Cohort 2: 2 mg ERX-963 Period
Number analyzed (Participants) | 7 | 7 | 5 | 5
score on a scale
  baseline Stanford Sleepiness Score | 3.4 (0.79) | 3.4 (0.79) | 4.0 (2.12) | 4.2 (2.17)
  10 min. after end of infusion, SSS | 3.0 (0.82) | 2.7 (1.60) | 4.0 (1.87) | 3.8 (2.39)
  40 min. after end of infusion, SSS | 3.1 (1.57) | 2.9 (1.68) | 4.2 (1.92) | 4.0 (2.45)
  1 hr., 10 min. after end of infusion, SSS | 3.7 (1.98) | 3.1 (1.57) | 4.0 (1.73) | 5.0 (2.45)
  1 hr., 40 min. after end of infusion, SSS | 3.6 (1.40) | 3.3 (0.76) | 4.6 (1.82) | 5.6 (1.82)
Statistical Analysis 1: Comparison: Cohort 1: Placebo Period vs Cohort 1: 1 mg ERX-963 Period vs Cohort 2: Placebo Period vs Cohort 2: 2 mg ERX-963 Period; A mixed effects model will be used to compare SSS effects following ERX-963 versus placebo. In the primary analysis of SSS, the cohort 1 and cohort 2 data were combined for ERX-963 and placebo treatments; Test type: Superiority; p = 0.7746, Mixed Models Analysis; mixed effects model = -0.0796, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.2768
Statistical Analysis 2: Comparison: Cohort 1: Placebo Period vs Cohort 1: 1 mg ERX-963 Period; A mixed effects model will be used to compare SSS effects following 1 mg ERX-963 versus placebo. In this analysis of SSS, the effect of 1 mg ERX-963 treatment was compared to the effect of placebo treatment; Test type: Superiority; p = 0.4700, Mixed Models Analysis; mixed effects model = -0.2608, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.3589
Statistical Analysis 3: Comparison: Cohort 2: Placebo Period vs Cohort 2: 2 mg ERX-963 Period; A mixed effects model will be used to compare SSS effects following 2 mg ERX-963 versus placebo. In this analysis of SSS, the effect of 2 mg ERX-963 treatment was compared to the effect of placebo treatment; Test type: Superiority; p = 0.8127, Mixed Models Analysis; mixed effects model = 0.1016, 95% CI 2-sided [-0.8 to 1.0], Standard Error of Mean 0.4272

3. Secondary Outcome: Assess the Effect of ERX-963 on the Change in Patient Global Impression - Improvement Scale (PGI-I) Compared to Placebo
Description: The PGI-I is a 7-point rating system used by the patient to rate their overall clinical condition after intervention relative to before intervention where 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse, and 7=very much worse.
Time Frame: Administered at the end of the dosing visit day, upon completion of the other outcome measures. Approximately 2 hours after the end of infusion.
Population: All treated participants who completed all the protocol specified assessments in both treatment periods were analyzed.
Measure: Mean (Standard Deviation); unit: Score of a scale
Groups:
- Cohort 1: 1 mg ERX-963 Period; Cohort 2: Placebo Period; Cohort 2: 2 mg ERX-963 Period: The crossover design tests each subject under different treatment conditions allowing for each subject to serve as their own control.
  Sequence 1: Participants will receive placebo followed by a washout period. After the washout period, participants will receive 2 mg of ERX-963.
  Sequence 2: Participants will receive 2 mg of ERX-963 followed by a washout period. After the washout period, participants will receive placebo.
Arm/Group | Cohort 1: Placebo Period | Cohort 1: 1 mg ERX-963 Period | Cohort 2: Placebo Period | Cohort 2: 2 mg ERX-963 Period
Number analyzed (Participants) | 7 | 7 | 5 | 5
Score of a scale | 3.4 (1.27) | 3.4 (1.13) | 4.0 (2.00) | 4.2 (1.92)

4. Secondary Outcome: Assess the Effect of ERX-963 on the Clinical Global Impressment - Improvement (CGI-I) Scale Compared to Placebo
Description: The CGI-I is a 7-point rating system used by the clinician or investigator to compare the patient's overall clinical condition after intervention relative to before intervention where 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse, and 7=very much worse (Guy, 1976; Busner, 2007).
Time Frame: as for outcome 3
Population: All treated participants who completed all the protocol specified assessments in both treatment periods were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo Period | Cohort 1: 1 mg ERX-963 Period | Cohort 2: Placebo Period | Cohort 2: 2 mg ERX-963 Period
Number analyzed (Participants) | 7 | 7 | 5 | 5
Score on a scale | 3.7 (1.25) | 3.9 (0.90) | 4.0 (1.22) | 4.4 (1.67)

5. Secondary Outcome: Assess the Effect of ERX-963 on the Psychomotor Vigilance Task (PVT)
Description: Participants will be tested for their response time and number of lapses during the PVT.
Time Frame: From dosing to approximately 2 hours
Population: PVT analysis was not performed for this study as this outcome measure analysis requirement was removed in the amended statistical plan. At the end of the clinical study, the project was terminated and the development group was disbanded. The entire team that worked on this project departed and moved on to their new companies. Therefore, this Outcome Measure has zero total analyzed.
Arm/Group | Cohort 1: 1 mg ERX-963 | Cohort 2: 2 mg ERX-963
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Assess the Effect of ERX-963 on the One-back Task
Description: Participants will be tested for the proportion of correct response to the One-back task.
Time Frame: From dosing to approximately 2 hours
Population: One-back task analysis was not performed for this study as this outcome measure analysis requirement was removed in the amended statistical plan. At the end of the clinical study, the project was terminated and the development group was disbanded. The entire team that worked on this project departed and moved on to their new companies. Therefore, this Outcome Measure has zero total analyzed.
Arm/Group | Cohort 1: 1 mg ERX-963 | Cohort 2: 2 mg ERX-963
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from screening to the End of Study Visit, which was a period of up to 57 days
Description: The adverse event and serious adverse event definition for this study did not differ from the clinicaltrials.gov definitions.
  Treatment-emergent AEs were AEs which started between the date and time of study drug dosing and through Study Day 2, within each period.
  Drug-related AEs were assessed by the investigator to determine the relationship (related or unrelated) between the study intervention and each AE occurrence.
Arm/Group | Cohort 1: Placebo Period | Cohort 1: 1 mg ERX-963 Period | Cohort 2: Placebo Period | Cohort 2: 2 mg ERX-963 Period
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 2/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo Period (N=7) | Cohort 1: 1 mg ERX-963 Period (N=7) | Cohort 2: Placebo Period (N=5) | Cohort 2: 2 mg ERX-963 Period (N=5)
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The 0.5 mg dose level was not tested in this study.

The analyses of the effect of ERX-963 on the Psychomotor Vigilance Task and the One-Back task were removed from the final analysis and documented accordingly in a Statistical Analysis Plan memo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Expansion Therapeutics reserves the right to embargo communications regarding trial results prior to public release for a period ≤ 60 days in order to protect patentable information. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed company confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT03959189/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT03959189/SAP_001.pdf